CLINICAL TRIAL: NCT03000985
Title: Evaluation of a Psychoeducation Program for Families Caregivers of Schizophrenic Patients : Randomized Study in Two Arms
Acronym: PSYEDUC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Charles Perrens, Bordeaux (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PHRIP PSY EDUC 2013
Record Dates: First submitted 2016-12-16; First posted 2016-12-22 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Schizophrenia; Mental Disorder; Educational Problems; Family Relations; Relapse; Medication Adherence; Psychiatric Disorder; Psychiatric Hospitalization
Keywords: schizophrenia; psychoeducation program; family caregiver; relapse; medication adherence; burden
MeSH Terms: conditions — Schizophrenia; Mental Disorders; Recurrence; Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducation (Experimental): 6 session of a psychoeducation program with the family. Psychoeducation focuses on explaining schizophrenia as a medical illness, the prognosis, and how the patient and family can increase the likelihood of better outcome.
  Interventions: Behavioral: Psychoeducation
- Control (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Psychoeducation — 6 session psychoeducation program with the family caregiver of schizophrenics patients.
  Arms: Psychoeducation

SUMMARY:
The involvement of family members is crucial and improves the prognosis of psychiatric patients and reinforces therapeutic adherence and reduces the frequency of relapses. For schizophrenia, the scientific literature clearly shows that it's in the interest of the patient to offer to his family a psychoeducational program.

Therapeutic education programs are now part of the recommendations of good clinical practice and in the French health through the law n ° 2009-879 of July 21, 2009 on the reform of the hospital and relating to patients, health and territories.

DETAILED DESCRIPTION:
Objectives We conducted a randomized study in two groups to evaluate the impact of a psychoeducational program for caregivers.

Methods 60 patients with a DSM-V diagnosis of schizophrenia and their families' caregivers are recruited. Families' caregivers are randomly assigned to receive either a 6 session psychoeducation program, or no psychoeducation.

Baseline evaluations:

Patients: symptomatology (PANSS), medication adherence (MARS); Families' Caregivers: Quality of Life (S-CGQoL), Burden (Zarit), knowledge of disease (KAST), therapeutic alliance (4PAS caregivers), depression (CES-D), medication adherence (CRS).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, based on ICD-10 (F20 to F29)
* Receive in-patient treatment at hospital (or medical center linked to Charles Perrens Hospital)
* Be the caregiver or parent of the patient
* Patient informed of the diagnosis of his disease

Exclusion Criteria:

* Mental retardation or other diagnoses that could affect the ability to answer questionnaires, after the acute schizophrenia psychosis is controlled
* Suicidal ideation
* Non-comprehension of the French language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Relapse | baseline (pre-treatment) to six months post-baseline
  Reduction in the rate of relapse (hospitalization) in patients whose family participated in the psychoeducation group compared to patients without psychoeducation.
Medication adherence (caregiver perception) | baseline (pre-treatment) to six months post-baseline.
  Change from baseline (pre-treatment) to 6 months post-baseline in caregiver-report of medication adherence using respectively the Compliance Rating Scale.

SECONDARY OUTCOMES:
Quality of Life | baseline (pre-treatment) to six months post-baseline
  Change from baseline (pre-treatment) to 6 months post-baseline in patient-report of quality of life using the Schizophrenia Caregiver Quality of Life questionnaire.
Burden | baseline (pre-treatment) to six months post-baseline
  Change from baseline (pre-treatment) at 6 months post-baseline in family-report of burden using the Zarit Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Charles PERRENS, Bordeaux, France

REFERENCES:
- [Background] Misdrahi D, Petit M, Blanc O, Bayle F, Llorca PM. The influence of therapeutic alliance and insight on medication adherence in schizophrenia. Nord J Psychiatry. 2012 Feb;66(1):49-54. doi: 10.3109/08039488.2011.598556. Epub 2011 Aug 10. PMID 21830849
- [Derived] Tessier A, Roger K, Gregoire A, Desnavailles P, Misdrahi D. Family psychoeducation to improve outcome in caregivers and patients with schizophrenia: a randomized clinical trial. Front Psychiatry. 2023 Jun 23;14:1171661. doi: 10.3389/fpsyt.2023.1171661. eCollection 2023. PMID 37426102